CLINICAL TRIAL: NCT05609604
Title: Role of Trans-cranial Direct Current Stimulation in Appetite and Weight Control: A Prospective Randomized Study
Brief Title: Role of Transcranial Direct Current Stimulation in Appetite and Weight Control
Acronym: TDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No trained/ qualified staff available to perform study.
Sponsor: University at Buffalo (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Paresh Dandona, SUNY Distinguished Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TDCS Weight Loss
Record Dates: First submitted 2017-01-31; First posted 2022-11-08 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss; Appetite Loss
Keywords: TDCS; Obesity; Appetite; Weight loss
MeSH Terms: conditions — Weight Loss; Anorexia; Obesity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- active tDCS (Active Comparator): This group will receive 30 minutes of active stimulation from tDCS
  Interventions: Device: tDCS
- sham tDCS (Placebo Comparator): This group will receive 30 minutes of sham (placebo) stimulation from tDCS
  Interventions: Device: Shame- No current

INTERVENTIONS:
Device: tDCS — Electric current will be delivered to the pre-frontal cortex for 30 minutes.
  Arms: active tDCS
Device: Shame- No current
  Other Names: No current control arm
  Arms: sham tDCS

SUMMARY:
To study the effects of transcranial direct current stimulation (tDCS) on weight and appetite.

DETAILED DESCRIPTION:
1. To compare weight loss over one month in active tDCS group with sham tDCS group. The investigator will measure weight of every participants at the beginning of the study and one month after the last session of tDCS
2. To compare change in insulin sensitivity over one month in active tDCS group with sham tDCS group. The investigator will measure fasting insulin and glucose level, and calculate homeostatic model assessment-insulin resistance (HOMA-IR)
3. To compare change in cognitive performance as a response to food over one month in active tDCS group with sham tDCS group. The investigator will evaluate performance in a computerized task that measures executive functions under the presence of food (working memory, inhibitory control and a combination of both). The investigator will assess changes in accuracy and speed in the task under active tDCS versus sham tDCS.
4. To compare change in post-prandial glucose excursion and average meal counts per day. The investigator will use continuous glucose monitor to record the frequency and amplitude of glucose excursion.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 80 years of age
* Body mass index > 30 kg/m2

Exclusion Criteria:

* Current participation in any other concurrent clinical trials or previous participation within 30 days before the screening visit
* Pregnancy or premenopausal women who are trying to be pregnant
* Patients who are incompetent to give consent
* Obesity due to a known secondary cause (Cushing's syndrome, hypothyroidism, etc) or a history of weight loss surgery
* Have taken any of the following medications within the past 3 months:

  * phentermine, naltrexone, bupropion, topiratmate, lorcaserin, phendimetrazine, methamphetamine, benzphetamine, diethylpropion
* Any contraindication to receive transcranial direct current stimulation (tDCS):

  * Personal or family history of seizures, epilepsy or other unexplained loss of consciousness.
  * Current or past history of skin disease or damaged skin on the scalp at the site of stimulation (i.e. eczema, skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.).
  * Prior neurosurgical procedure or radiation.
  * Known diagnosis of brain lesions, such as tumor, stroke or multiple sclerosis
  * Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, Transcutaneous Electrical Nerve Stimulation unit, ventriculo-peritoneal shunt or any metallic implant on the head.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS: This group will receive 30 minutes of sham (placebo) stimulation from tDCS
  Shame- No current
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (3) | 43 (5) | 45 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 41 (5) | 38 (4) | 39.7 (4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: change in body weight in Kg measured from baseline at 5 weeks
Time Frame: 5 weeks
Population: no patient completed the study due to study termination due to departure of trained staff.
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05609604/Prot_SAP_000.pdf